CLINICAL TRIAL: NCT03728322
Title: A Safety and Efficacy Study of a Single Center, Open-label, Single Arm About the Gene Correction of HBB in Patient-specific iHSCs Using CRISPR/Cas9 That Intervent Subjests With β-thalassemia Mutations
Brief Title: iHSCs With the Gene Correction of HBB Intervent Subjests With β-thalassemia Mutations
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Allife Medical Science and Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HBB HSC-01
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-10

CONDITIONS: Thalassemia
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iHSCs treatment group (Experimental)
  Interventions: Biological: iHSCs treatment group

INTERVENTIONS:
Biological: iHSCs treatment group — iHSCs intravenous injection

SUMMARY:
This is a single centre、single arm、open-label study，to investigate the safety and efficacy of the gene correction of HBB in patient-specific iHSCs using CRISPR/Cas9.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of transplantation iHSCs intervent subjests with β-thalassemia mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 2 and ≤ 60 years of age
2. Subjects was confirmed the transfusion-dependent β-thalassemia
3. Adequate organ function, as defined by:

   Serum creatinine ≤ 1.5 mg/dl ； Serum ALT/AST）≤2.5×ULN；ALB≥25g/L； Serum total bilirubin < 1.5x ULN Left ventricular ejection fraction≥50%
4. Chest X-ray and ecg test results were normal, no serious cardiopulmonary diseases
5. Subjects survival was expected≥6 months
6. Adult patients were willing to use reliable contraceptives (such as condoms) and not to donate sperm throughout the study period and within three months of discharge
7. Subjects and the guardians able to undergo post-physical therapy/rehabilitation

Exclusion Criteria:

1. Subjects allergic to macromolecular biological agents such as antibodies or cytokines
2. Subjects receipt of any investigational clinical trials within 3 months.
3. Subjects previous treatment with any hematopoietic stem cell transplantation or other organ transplantation
4. Uncontrolled bleeding symptoms
5. Severe cardiovascular disease is known, including any of the following:

   Myocardial infarction or thrombosis has occurred in the past six months Subjects with unstable angina pectoris Subjects with Class III/IV cardiovascular disability according to the New York Heart Association Classification
6. Subjects have one kinds of tumors within 5 years
7. Active hepatitis B (HBV DNA>1000copy/mL), hepatitis C or HIV infection.
8. Subjects have an infectious diseases that cannot be controlled within 4 weeks
9. subjects have severe central nervous system disease or epilepsy
10. Subjects are Suffering from mental illness; Patients with alcohol dependence, drug abuse, drug addiction, and medical, psychological or social conditions that may interfere with research or have an impact on the evaluation of research results
11. Women in pregnancy (positive urine/blood pregnancy test) or lactation
12. Subjects who have other conditions that were not appropriate for the group determined by the researchers.

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment related adverse events as assessed by CTCAE v4.0 | 1 year
  Defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment